CLINICAL TRIAL: NCT06497673
Title: Sanger Human Cell Atlasing Project. Defining Human Cells in Terms of Gene Expression, Physiological States,Developmental Trajectories, and Location.
Brief Title: Sanger Human Cell Atlasing Project
Acronym: HCA
Status: Enrolling by invitation | Type: Observational
Sponsor: The Wellcome Sanger Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 260474
Record Dates: First submitted 2024-07-04; First posted 2024-07-12 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Human Development; Genetic Disease
MeSH Terms: conditions — Genetic Diseases, Inborn | interventions — Specimen Handling

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Samples will include whole or dissected tissues, frozen or fixed samples, single cell suspension and/or purified nucleic acids. Peripheral blood mononuclear cells (PBMCs), primary human umbilical vein endothelial cells (HUVEC), whole blood, bone marrow, urine, tissue samples and cell lines. Fetal samples will be received up to 24 weeks post conception.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: sample collection — New collected samples, as well as surplus surgical and diagnostic samples.

SUMMARY:
"Cell Atlasing" refers to a novel strategy to characterise cells in tissues at the molecular level in a quantitative manner. The international Human Cell Atlas consortium brings together a community of biologists, clinicians, technologists, physicists, computational scientists, software engineers, and mathematicians to capitalise on drawing together leaders with various biological, technical and computational expertise. The project is based on the aim to define all human cell types in terms of their distinctive patterns of gene expression, physiological states, developmental trajectories, and location. This will pave the way to create a reference map of all human cells as a basis for understanding human health and diagnosing, monitoring, and treating disease.

DETAILED DESCRIPTION:
Previous methods for quantifying molecular states of cells included microarray and standard RNA-seq analysis on a tissue section (RNA-seq is a technique to look at the activity of all the genes in a cell). These methods estimate the activity of any given gene by averaging the signal from millions of cells. Given the heterogeneity of cell populations (i.e.how uniform they are), measurement of the mean values of signals overlooks the internal interactions and differences within a cell population that may be crucial for maintaining normal tissue function and facilitating disease progression.

The Sanger Human Cell Atlasing project will adopt various genomic approaches that will provide genome-wide information in a single experiment. This project aims to scale up the single cell genomics and high-throughput highly multiplex spatial gene expression profiling approaches. Coupled with powerful computational methods, this strategy will produce a comprehensive and systematic reference map of human cells, providing a fundamental blueprint of cell states for both basic biological research and clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Samples are from the living and the deceased age 0 to 99+ from healthy and diseased individuals.
* All samples will have fully informed consent for use in research.

Exclusion Criteria:

* Samples taken without consent for use in future research
* Samples taken from individuals without the capacity to consent to use in research

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Samples are from the living and the deceased age 0 to 99+ from healthy and diseased individuals, to facilitate atlasing of the entire human body.
  Samples for this study will be obtained from tissue banks and ethically approved research studies where consent has been taken for use of the samples in future research.
  Prospective samples will also be collected via collaborators at NHS sites. This will allow for the collection of all cell types to fulfil the aims of the study. We will provide collaborators with study specific participant information sheets and informed consent forms to recruit potential donors.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2019-12-16 (Actual); Primary Completion 2029-11-07 (Estimated); Study Completion 2029-11-07 (Estimated)

PRIMARY OUTCOMES:
This project aims to scale up the single cell genomics and high-throughput highly multiplex spatial gene expression profiling approaches. | 10 years
  Coupled with powerful computational methods, this strategy will produce a comprehensive and systematic reference map of human cells, providing a fundamental blueprint of cell states for both basic biological research and clinical practice.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Teichmann, Principal Investigator — Wellcome Sanger Institute
Locations (1):
- Wellcome Sanger Institute, Cambridge, United Kingdom